CLINICAL TRIAL: NCT01086098
Title: Trends in Cardiac Pacing - 30 Years of Implants
Brief Title: PACE30: 30 Years in Cardiac Pacing
Acronym: PACE30
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, AChoy, Consultant, University of Dundee
Other Study IDs: ELD004
Record Dates: First submitted 2010-03-05; First posted 2010-03-12 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2010-03

CONDITIONS: Pacemakers
Keywords: Pacemakers; Survival

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All paced patients

SUMMARY:
Limited data exist regarding temporal trends in permanent pacemaker (PPM) implantation. To describe trends in incidence and comorbidities of PPM recipients, the investigators aim to conduct a retrospective population-based cohort study using record linkage, over a 32 year period.

ELIGIBILITY:
Inclusion Criteria:

* All patients with pacemakers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with pacemakers
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2010-03-01 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2011-03-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Mortality | 30 years
  We will examine time to cardiovascular death from pacemaker implant and relate to the differing indications for pacing

SECONDARY OUTCOMES:
Hospitalisation for heart failure | 30 years
  We will examine the frequency of hospitalisations after device implantation